CLINICAL TRIAL: NCT06605053
Title: ENding HIV Transmission to Infants by Generating Evidence to Optimize Prevention and Care for Pregnant and Postpartum Adolescent Girls and Young Women With HIV in Tanzania (ENGAGE)
Brief Title: Optimizing Prevention and Care for Pregnant and Postpartum Adolescent Girls and Young Women With HIV in Tanzania
Acronym: ENGAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Management and Development for Health, Tanzania (Unknown)
Responsible Party: Principal Investigator, Anna Kågesten, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-00911; NIMR/HQ/R.8a/Vol.IX/4637 (Other: Tanzania National Institute for Medical Research)
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: HIV Antiretroviral Therapy (ART) Adherence; PMTCT; Pregnancy; Retention in Care; HIV Viremia; Early Infant HIV Diagnosis
Keywords: Adolescent girls and young women; HIV; Vertical transmission; PMTCT; Co-production; Co-design; Intervention; Tanzania; Sub-Saharan Africa; Retention in care

STUDY DESIGN:
Intervention Model Description: A two-arm, cluster randomized implementation trial in routine healthcare settings providing day-to-day vertical HIV prevention services in Dar es Salaam (urban) and Kagera (rural) regions of Tanzania to pilot test a co-produced intervention package for feasibility, acceptability, and preliminary effect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (co-produced intervention package to optimize PMTCT care) (Experimental): Pregnant girls/young women 15-24 years living with HIV (new, previously diagnosed, and transfers) receiving PMTCT services in routine healthcare randomized to the intervention between 01st January and 30th June 2026 and followed up for at least one year to 30th June 2027. While the specific intervention will developed earlier in the project, it may include a package of evidence-based approaches such as peer mentor mothers, male partner involvement, flexible hours for girls/young women and mobile phone reminders. A focal team of 2-3 persons will be trained and engaged to drive the implementation of the interventions at randomized faciltiies. The focal team will orient and engage other staff and stakeholders to deliver the interventions, identify and address gaps, and monitor implementation fidelity and quality using standard operating procedures.
  Interventions: Behavioral: Co-produced intervention to optimize PMTCT care engagement
- Control: standard care (No Intervention): Pregnant AGYW living with HIV (new, previously diagnosed, and transfers) receiving vertical HIV prevention services in routine healthcare centres acting as control facilities, between 01st January and 30th June 2026 and followed up for at least one year to 30th June 2027. No intervention is administered to this arm; participants will receive a standard of care for PMTCT services per Tanzania national guidelines.

INTERVENTIONS:
Behavioral: Co-produced intervention to optimize PMTCT care engagement — While the specific interventions package will developed earlier in the project, it may include evidence-based approaches such as peer mentor mothers, male partner involvement, flexible hours for girls/young women and mobile phone reminders. Overall, the interventions should be brief and easy to integrate into standard care, aiming to 'nudge' or motivate participants (towards improved engagement, retention, and outcomes) as well as health care providers or community stakeholders to better understand and support girls/young women's specific needs. A focal team of 2-3 persons will be trained and engaged to drive the implementation of the interventions at randomized faciltiies. The focal team will orient and engage other staff and stakeholders to deliver the interventions, identify and address gaps, and monitor implementation fidelity and quality using standard operating procedures.
  Arms: Intervention arm (co-produced intervention package to optimize PMTCT care)

SUMMARY:
The goal of this clinical trial is to find better ways to care for pregnant and postpartum adolescent girls and young women (AGYW) aged 15-24 years with HIV in Tanzania, and to prevent them from passing HIV to their babies. The main questions it aims to answer are:

* How often do young pregnant women with HIV go to their health appointments and stay on their treatment up to two years after giving birth?
* How many babies born to young women with HIV stay HIV-free for two years?
* How soon do young women with HIV get pregnant again after giving birth, and what factors affect this?
* What are the best ways to help young women with HIV stay in care and stay healthy during and after pregnancy?
* What social and structural factors affect whether young pregnant women with HIV go to their health appointments and stay on their treatment?
* How can we work with young women with HIV to create and test a package of interventions to improve their healthcare during and after pregnancy?
* Can this package of interventions help young women with HIV stay in care and remain healthy during and after pregnancy?

Participants will:

* Have their health data analyzed via health service records of all women who received HIV prevention services between 2018 and 2020, and were followed until 2023, across 559 health facilities in Tanzania.
* Participate in qualitative interviews to share their experiences and challenges with staying in care.
* Help to co-create a package of interventions to improve care.
* Take part in a cluster-randomized trial to test these interventions. Researchers will compare the outcomes of the intervention package to see if they improve care engagement, retention, and health outcomes for AGYW with HIV during and after pregnancy.

DETAILED DESCRIPTION:
Background Sub-Saharan Africa (SSA) remains the most affected region by the global HIV pandemic, accounting for half of all new HIV infections and 66% of the world's 39 million people living with HIV (PLHIV). In SSA, two-thirds of new HIV infections occur among women of reproductive age, with adolescent girls and young women (AGYW) aged 15-24 years being 3.5 times more likely to acquire HIV compared to young men. Pregnant AGYW with HIV face poorer outcomes on antiretroviral treatment (ART) and have elevated risks of vertical HIV transmission to their infants.

In 2022, SSA had 84% of the 130,000 estimated new HIV infections in children aged 0-14 years globally, with vertical transmission accounting for over 90% of these cases. Effective use of ART among pregnant and breastfeeding women with HIV can reduce the risk of vertical HIV transmission to less than 2%. However, significant gaps remain, with Tanzania being one of the countries with the highest numbers of new HIV infections in children and women of reproductive age. Despite progress in reducing vertical transmission rates, pregnant AGYW continue to lag in efforts to end HIV infections in children, having poorer HIV treatment outcomes, higher vertical transmission rates, and higher reproductive health risks. While good quality evidence on AGYW is missing; available data shows that AGYWs' specific needs are not sufficiently addressed by standard care. There is, therefore, an urgent need to expand knowledge on and explore effective approaches to improve HIV and reproductive healthcare experience and outcomes for pregnant AGYW with HIV.

Study Objectives The purpose of the ENGAGE project is to optimize care for prevention of vertical HIV transmission and HIV treatment among pregnant and postpartum AGYW with HIV and their infants, and to improve the prevention of unintended pregnancies among AGYW in Tanzania - a setting where HIV is endemic and maternal mortality remains a leading cause of death among young women.

This is done via four sub-studies with the following specific objectives:

Sub-study 1:

* To investigate patterns and trends of health service uptake, retention and health outcomes among pregnant/ postpartum AGYW living with HIV up to two years after delivery.
* To determine 2-years HIV-free survival rate among infants born to AGYW living with HIV.
* To assess the timing and spacing of subsequent pregnancies, and factors influencing them, among AGYW living with HIV enrolled in prevention of vertical HIV transmission services.

Sub-study 2:

* To synthesize available evidence on potential interventions to improve health service uptake, retention and health outcomes among pregnant/ postpartum AGYW living with HIV enrolled in prevention of vertical HIV transmission services.
* To understand social-structural factors influencing health service uptake, retention and health outcomes among pregnant/ postpartum AGYW living with HIV.

Sub-study 3:

• To co-create and prototype a tailored package of micro-interventions to optimize healthcare for prevention of vertical HIV transmission services for AGYW.

Sub-study 4:

• To assess the feasibility and preliminary effect of a micro-intervention package tailored to improve service uptake, retention and health outcomes among pregnant AGYW living with HIV.

Study Design and setting This is a mixed-methods implementation research project embedded within routine healthcare settings. It employs a sequential explanatory design, starting with an analysis of quantitative cohort data on adolescent girls and young women (AGYW) enrolled in PMTCT Option B+ (sub-study 1). This is followed by a stepwise qualitative inquiry aimed at co-producing and prototyping a package of interventions that can be seamlessly integrated to enhance existing care approaches (sub-studies 2-3). The intervention package will then be pilot-tested for feasibility and preliminary effectiveness using a cluster-randomized clinical trial design (sub-study 4).

The project will be conducted in the regions of Dar es Salaam, Kagera, and Tabora in Tanzania. Dar es Salaam, the most populous and main commercial hub of Tanzania, is predominantly urban with a population of 5.4 million out of the country's 62 million. In contrast, Kagera and Tabora are primarily rural, with populations of 3.0 million and 3.4 million, respectively. The prevalence of HIV among adults aged 15 and older is 4.2% in Dar es Salaam, 5.7% in Kagera, and 5.6% in Tabora. Annually, these regions see approximately 200,000 new pregnant women attending antenatal care (ANC) clinics in Dar es Salaam, 140,000 in Kagera, and 200,000 in Tabora, with 3%-4% of these women being HIV positive. Among these HIV-positive pregnant women, those aged 15 to 24 years constitute about 20% in Dar es Salaam, 27% in Kagera, and 24% in Tabora.

Sub-study I: Registry-based Retrospective Cohort Design and Participants: This observational cohort study utilizes data from routine healthcare records of 559 MDH-supported health facilities, which account for over 90% of HIV care in the three regions of Dar es Salaam, Kagera, and Tabora. The study includes all pregnant/postpartum AGYW with HIV who started vertical HIV prevention services between January 1, 2018, and December 31, 2020, and their infants born from this pregnancy/breastfeeding episode.

Data Collection and Analysis: Data will be sourced from the Tanzania national electronic CTC2 database, which stores information on HIV care and vertical HIV prevention services. The primary outcomes measured include time to ART attrition, detectable viral load, and HIV-free infant survival. Secondary outcomes include repeat pregnancy, uptake of vertical HIV prevention services, and maternal/pregnancy loss. Data will be analyzed using statistical methods such as the Kaplan Meier method, Cox regression, generalized estimating equations (GEE), and Poisson regression.

Limitations and Mitigation: The study acknowledges challenges related to the quality and completeness of routinely collected data. To address these issues, physical verification will be performed by obtaining patient charts and updating the CTC2 database. Multiple methods, including multiple imputation and propensity scores, will be employed to handle incomplete or missing data.

Sub-study II: Evidence Review and Consultations Part 1: Evidence Review Design and Scope: A systematic review based on the PRISMA guidelines will be conducted to identify potential interventions to improve engagement, retention, and health outcomes of vertical HIV prevention services among AGYW in SSA. The review will include experimental designs with a control group and will focus on studies conducted between 2014 and 2023.

Search Strategy and Data Extraction: Peer-reviewed articles and grey literature will be searched using databases such as PubMed and Medline. The search strategy will consider the four PICO elements (Patient/Population/Problem, Intervention, Comparison, and Outcomes) to develop the search syntax. Data extraction will be done using a standardized excel sheet to capture key study aspects.

Synthesis and Risk of Bias Assessment: For experimental studies, meta-analysis will be conducted if feasible. Otherwise, findings will be synthesized using a comprehensive narrative approach. Risk of bias will be assessed using appropriate tools for each study type, and the overall certainty of evidence will be rated using the Cochrane GRADE approach.

Part 2: Qualitative consultations will be conducted through in-depth interviews (IDIs) and focus group discussions (FGDs) with AGYW ages 15-24 years, healthcare providers, spouses/partners, parents, and community stakeholders. The study will be conducted in Dar es Salaam (urban) and Kagera (rural) regions.

Data Collection and Analysis: Participants will be recruited using purposive sampling. Data will be collected using semi-structured interview guides and analyzed using content analysis. Themes and subthemes will be identified and discussed by the research team.

Sub-study III: Co-design and Prototyping of an Intervention package Design and Participants: This stage involves co-creating a package of interventions with AGYW, healthcare providers, and community stakeholders. The participants will be organized into an intervention development group consisting of about 24 members, including pregnant and postpartum AGYW, spouses/partners, parents/guardians, healthcare providers, community stakeholders, and research team members.

Co-production Process: The co-production process will be conducted through a series of workshops over six months. The workshops will be held in neutral, accessible, and safe community/public venues to enhance active interactions. Participants will use various methods of participation, including flash cards, role play, and writing on whiteboards/flip charts/sticky notes. The outcome will be a package of interventions designed to improve engagement, retention, and outcomes of AGYW in vertical HIV prevention services.

Prototyping Stage: During the prototyping stage, the intervention development group, research team, and other reproductive health/AGYW experts will draft intervention materials and training manuals. These will be tested at 1-2 purposefully selected intervention facilities. The process will involve training healthcare providers or other stakeholders to deliver the interventions and gaining input from AGYW and providers on the acceptability of the content and methods.

Sub-study IV: Pilot-test the Intervention Package Design and Participants: two-arm cluster randomized trial to evaluate the feasibility, acceptability, and preliminary effectiveness of the interventions in Dar es Salaam and Kagera regions of Tanzania. Participants will include pregnant AGYW living with HIV (new, previously diagnosed, and transfers) who are receiving vertical HIV prevention services between January 1, 2026, and June 30, 2026, with follow-up extending for at least one year until June 30, 2027.

Sampling Method and Sample Size: The sample size for the study was estimated using a formula for cluster randomized studies, which inflates the sample size for a two-arm simple randomized study using the design effect. The design effect accounts for the clustering effect with an intra-cluster correlation coefficient (ICC) of 0.02 and an average cluster size of 12. The final sample size is determined to be 222 participants (111 per arm), providing 80% power to detect a 15% difference in retention rate between the intervention and control arms with a standard error of 0.05.

Facility Sampling and Randomization: Between 2018 and 2020, 376 MDH-supported facilities provided vertical HIV prevention services to at least one AGYW in Dar es Salaam and Kagera regions. From these, 225 facilities that enrolled at least 10 AGYW per year were identified: 116 in Dar es Salaam and 139 in Kagera. The facilities include hospitals, health centers, and dispensaries. Using block randomization, 12 facilities per region will be randomized into six intervention and six control arms, ensuring a balanced distribution of facility levels.

Intervention and Control: At each intervention facility, a focal team of 2-3 persons, comprising both AGYW and healthcare providers, will be trained and engaged to drive the implementation of the intervention package. This team will orient and engage other staff and stakeholders to deliver the interventions, identify and address gaps, and monitor implementation fidelity and quality using standard operating procedures and job aids. The interventions will be integrated into routine care, with hands-on supportive supervision and mentorship provided by local researchers through weekly follow-ups in the first month and monthly thereafter. The intervention package may include components such as SMS/phone call reminders, peer mother support, and flexible clinic hours tailored to the needs of AGYW. The control arm will received standard PMTCT care as per national Tanzania guidelines.

Data Collection and Analysis: Data for assessing the preliminary effect on primary outcomes will be extracted from the existing Tanzania national electronic CTC2 database. Data will be analyzed using statistical methods such as Kaplan Meier and Cox regression for time to ART attrition and HIV-free infant survival, generalized estimating equations (GEE) for detectable viral load, and Poisson regression for the composite outcome of optimal vertical HIV prevention. Additional qualitative data will be collected from AGYW and healthcare providers through face-to-face interviews using a semi-structured questionnaire.

Fidelity Assessment and Feasibility: To ensure comprehensive fidelity measurement, the study will use a combination of methods at various levels of implementation. These methods will include checklists, adherence reports, structured audits, and fidelity assessment protocols. Fidelity assessments will be conducted at baseline (before implementation begins), periodically (at weekly/monthly intervals during the intervention's implementation), and at the end of the intervention to evaluate overall fidelity.

Study Limitations and Mitigation: To address potential data quality issues in the CTC2 database, the study will implement rigorous validation and cleaning processes, cross-referencing with other sources, conducting data quality assessments, and addressing missing data through appropriate imputation methods. This approach aims to enhance the reliability and integrity of the study findings.

Ethical considerations The project has received ethical approval from the National Health Research Ethics Committee (NaTHREC) in Tanzania. Approval will also be sought from the Swedish Ethical Review Authority (EPM) for analysis of de-identified data in Sweden.

Key ethical aspects include:

* Informed Consent: Informed consent will be obtained from all participants involved in new data collection. For minors aged 15-17 years, who are considered emancipated, consent will be sought directly from them without the need for parental consent.
* Privacy and Confidentiality: The study involves the collection of sensitive personal information. To protect participants' privacy, personal identifiers such as names and addresses will not be extracted from the registry. Interviews will be conducted in pre-arranged, private spaces, and all study data will be stored securely in password-protected computers with access limited to the research team.
* Minimizing Risks: The study is designed to use routine healthcare data, supplemented by qualitative data from focus group discussions and interviews. The risks to participants are considered minimal, but potential risks and ethical considerations have been identified and addressed.

Implications The ENGAGE study represents a significant effort to address the unique needs of young women living with HIV in Tanzania, aiming to improve their health outcomes and reduce the risk of HIV transmission to their infants. Through a collaborative and evidence-based approach, the study seeks to contribute to the global goal of eliminating HIV/AIDS.

ELIGIBILITY:
Sub-study 1 (registry-based cohort analysis):

Inclusion Criteria:

* Pregnant/postpartum adolescent girls and young women (AGYW) with HIV aged 15-24 years, who started PMTCT services between January 1, 2018, and December 31, 2020.
* Infants born to the included AGYW during this period.

Exclusion Criteria:

* AGYW whose ART (Antiretroviral Therapy) status was not recorded.
* Women who had not started ART.

Sub-study 2 (qualitative):

Inclusion Criteria:

* AGYW living with HIV who are currently pregnant, previously pregnant/postpartum, and never pregnant).
* HCPs (Health Care Providers) at clinics providing PMTCT services.
* Spouses/partners/parents of AGYW and community stakeholders within the study setting.

Exclusion criteria

- Mentally or severely ill individuals unable to participate in the study activities.

Sub-study 3 (co-production)

Inclusion criteria:

* AGYW, HCPs, spouses/partners, parents, and community stakeholders who participated in the qualitative study II.
* Research team members.

Exclusion criteria:

- Mentally or severely ill individuals unable to participate in the study activities.

Sub-study 4 (cluster-randomized implementation trial)

Inclusion criteria:

- Pregnant AGYW living with HIV (new, previously diagnosed, and transfers) receiving vertical HIV prevention services in routine healthcare between January 1, 2026, and June 30, 2026, and followed up for at least one year until June 30, 2027.

Exclusion criteria:

* AGYW whose ART (Antiretroviral Therapy) status was not recorded.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time to ART attrition | 24 months
  The hazard rate of discontinuing ART for any reason including death, stopping ART or loss to follow-up for 90 consecutive days from scheduled appointment
Detectable viral load | 24 months
  The proportion of participants with detectable viral load, defined as ≥50 viral copies/mL of blood after at least three months of ART use (for those who started ART at enrolment) or detectable VL after enrolment (for those already on ART at enrolment).
HIV-free infant survival | 24 months
  Defined as the proportion of infant who are alive and tested negative at final HIV test by 18+ months postpartum, or last available data point

SECONDARY OUTCOMES:
Repeat pregnancy | 24 months
  Defined as the number of subsequent pregnancies occurring after the index pregnancy (at PMTCT enrolment) during the two years of post-partum follow-up period
Uptake of PMTCT services | 24 months
  Rate of uptake of PMTCT services in-line with national PMTCT guidelines, defined as (in relation to the index pregnancy): starting ART before/within the first trimester, making at least 8 visits before delivery, and receiving first infant HIV testing within 2 months postpartum.
Maternal/pregnancy loss | 24 months
  The proportion of participants ending in a maternal or pregnancy loss in relation to the index pregnancy, defined as miscarriage, stillbirth or maternal death.

OTHER OUTCOMES:
Acceptability | 24 months
  Qualitative themes related to acceptability of the intervention, based on thematic analysis of qualitative data from individual interviews with participants
Intervention feasibility | 24 months
  Qualitative themes related to feasibility of the intervention based on qualitative data collected during individual interviews

CONTACTS AND LOCATIONS:
Locations (2):
- Tanzania (2):
  - Management and Development for Health, Dar es Salaam
  - Management and Development for Health, Kagera

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data from the registry-based cohort will be available upon request, as a de-identified file. Primary participant data from qualitative interviews will not be shared outside of the research team in order to ensure the confidentiality and privacy of participants. A complete list of codes and themes from the qualitative analysis will be shared as part of publications.

REFERENCES:
- [Background] Lyatuu GW, Urrio R, Naburi H, Lyaruu P, Simba B, Siril H, Philipo E, Machumi L, Kibao A, Kajoka D, Nyamhagatta M, Sando D, Biberfeld G, Orsini N, Kilewo C, Ekstrom AM. Vertical HIV transmission within 18 months post partum among women on lifelong antiretroviral therapy for HIV in Dar es Salaam, Tanzania: a prospective cohort study. Lancet HIV. 2023 Jan;10(1):e33-e41. doi: 10.1016/S2352-3018(22)00289-2. Epub 2022 Dec 7. PMID 36495896